CLINICAL TRIAL: NCT01415362
Title: Development of a Closed-loop Detect-and-treat System Using Transcranial Direct Current Stimulation (tDCS) for Epilepsy
Brief Title: Closed-loop System Using Transcranial Direct Current Stimulation (tDCS) for Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2010-p-000289
Record Dates: First submitted 2011-07-26; First posted 2011-08-11 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Epilepsy; Seizures
Keywords: transcranial direct current stimulation; electroencephalography
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): The subject will receive sessions of active tDCS remotely triggered by the EEG monitoring system each time seizure activity is detected during the 24-hour period.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): The subject will receive sessions of sham tDCS remotely triggered by the EEG monitoring system each time seizure activity is detected during the 24-hour period.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — For both active and sham tDCS, the device will be hooked up to the closed loop system, using electrodes of 35cm^2. During active tDCS, the subject will receive 2mA for 5 min. During sham tDCS, the current will only be active for 30 seconds (current ramping up and then down) to simulate the sensations of active tDCS.
  The subject will undergo either active or sham stimulation for their first 24-hour EEG monitoring visit, and the opposite intervention on the second 24-hour EEG monitoring visit.
  Other Names: low intensity 1x1 direct current stimulator

SUMMARY:
In this pilot study, the researchers investigated the feasibility of a closed-loop electroencephalography (EEG) / transcranial direct current stimulation (tDCS) system for treatment of epilepsy. They looked to see the feasibility of triggering tDCS stimulation within 10 seconds of a detected EEG partial-onset seizure, and also a proof-of-principle determination of whether tDCS applied during this vulnerable period may be feasible to prevent the oncoming seizure.

This study required 5 visits over the course of approximately 8 weeks. Each visit was separated by at least 2 weeks. Two of the visits had 24-hour EEG monitoring sessions. During these two sessions, the EEG and tDCS were hooked into a closed loop system, such that when seizure activity wasdetected, the tDCS was triggered to deliver stimulation. Subjects received active stimulation or sham stimulation sessions during the first 24-hour visit, and the opposite during the second. The subjects were randomized and counterbalanced.

We have also added a healthy subjects cohort to assess the feasibility of the closed loop system. In order to test the proof-of-concept of this system, the experiment will focus on detecting and acting upon alpha- and beta-band changes traced in the EEG activity that is being recorded, and provide tDCS stimulation based upon those changes. We will enroll 6 subjects who will have 2 visits each. During these two visits subjects will be randomized to active or sham stimulation sessions and receive the opposite during their second visit.

ELIGIBILITY:
Inclusion Criteria (Epileptics)

* Disabling motor simple partial seizures, complex partial seizures, and/or secondarily generalized seizures. Disabling refers to seizures that are severe enough to significantly impair functional abilities in areas such as employment, psychological or social wellbeing, education or mobility.
* Failed treatment with a minimum of two antiepileptic medications.
* Experienced an average of three or more disabling simple weekly partial seizures, complex partial seizures and/or secondarily generalized seizures.
* Between the ages of 18 and 70 years.
* No more than two epileptogenic regions in the brain.
* Must be able to provide informed consent themselves.

Exclusion Criteria

* Has a progressive neurological or systemic disease.
* Has a history of nonepileptic seizures.
* Has an implanted metallic device, aneurysm clips, cochlear implants, or spinal cord stimulator.
* Has suffered a severe traumatic brain injury with skull fracture.
* Contraindications to tDCS

  * metal in the head
  * implanted brain medical devices
* Pregnancy
* Any implanted electrical medical device, including pacers and implanted cardiac defibrillators

Inclusion criteria (Healthy Subjects)

- Healthy subjects age 18 and older

Exclusion criteria:

* Existence of major neurologic or psychiatric condition (i.e. epilepsy, severe depression)
* History of head injury resulting in more than a momentary loss of consciousness
* Previous neurosurgery
* A history of significant alcohol or drug abuse in the prior 6 months
* Presence of unstable medical conditions, such as; uncontrolled diabetes mellitus, cardiac pathology, cancer, kidney insufficiency, acute thrombosis
* Contraindication to tDCS

  * metal in the head
  * implanted electronic medical devices
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Measurement of seizure activity via electroencephalography (EEG) | Measured for approximately 48 hours
  Measurement of seizure activity will take place in two visits of 24-hour seizure monitoring. During these visits, the EEG will record seizure information including (1) number of seizures, (2) severity of seizures, and (3) latency of seizures between sessions of stimulation.

SECONDARY OUTCOMES:
Subject self-report of seizure activity | Measured for approximately 8 weeks.
  Subject will keep a diary to monitor baseline seizure activity between study visits. This will be measured daily for the 8 weeks the subject will participate.
Measurement of healthy subjects EEG changes | Measured for approximately 2 hours
  We will compare changes in EEG from before stimulation to after stimulation in a healthy cohort. We will test the system to trigger in healthy subjects when there is an increase of beta frequency power and decrease of alpha frequency power. We will also assess whether the tDCS stimulation will return the background EEG rhythm toward a baseline pattern (increasing alpha, decreasing beta)
N-back memory and attention test | Measured for approximately 2 hours
  We will assess working memory and attention in healthy individuals using the n-back test, assessing changes from pre- to post-tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital (SRH)
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States